CLINICAL TRIAL: NCT03065647
Title: Extracorporeal CPR for Refractory Out-of-Hospital Cardiac Arrest (EROCA)
Brief Title: ECPR for Refractory Out-Of-Hospital Cardiac Arrest
Acronym: EROCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Food and Drug Administration (FDA) (U.S. Federal Agency); Physio-Control (Industry)
Responsible Party: Principal Investigator, Robert Neumar, Professor and Chair, Department of Emergency Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00117553; R34HL130738-01A1 (NIH)
Record Dates: First submitted 2017-02-16; First posted 2017-02-28 (Actual); Results first posted 2021-03-15 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Cardiac Arrest; Heart Arrest; Sudden Cardiac Arrest; Cardiopulmonary Arrest; Death, Sudden, Cardiac; Cardiopulmonary Resuscitation; CPR; Extracorporeal Cardiopulmonary Resuscitation; Extracorporeal Membrane Oxygenation
Keywords: Out-of-hospital cardiac arrest; Cardiac Arrest; Heart Arrest; Sudden Cardiac Arrest; Cardiopulmonary Resuscitation; Extracorporeal Cardiopulmonary Resuscitation; Extracorporeal Membrane Oxygenation; CPR; ECPR; ECMO; Emergency Medical Services; EMS; OHCA
MeSH Terms: conditions — Heart Arrest; Death, Sudden, Cardiac; Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Standard Care (No Intervention): Basic Life Support (BLS) and Advanced Cardiovascular Life Support (ACLS) by Emergency Medical Services (EMS) per existing EMS protocols at the scene of the cardiac arrest.
- Expedited Transport (Experimental): Intervention: Expedited Transport with Mechanical CPR.
  After initial Basic Life Support (BLS) and Advanced Cardiovascular Life Support (ACLS) by Emergency Medical Services (EMS) per existing EMS protocols, patients with refractory cardiac arrest are transported to an ECPR capable emergency department with ongoing mechanical CPR and ACLS for possible initiation of extracorporeal cardiopulmonary resuscitation (ECPR).
  Interventions: Device: Expedited Transport With Mechanical CPR

INTERVENTIONS:
Device: Expedited Transport With Mechanical CPR — Patients with OHCA refractory to initial BLS and ACLS will be transported by EMS with ongoing mechanical CPR and ACLS to an emergency department capable of initiating ECPR.
  Arms: Expedited Transport

SUMMARY:
In the U.S. alone, over 300,000 people per year have sudden out-of-hospital cardiac arrest (OHCA), and less than 1 out of 10 survive. The current standard practice for treating OHCA is to perform cardiopulmonary resuscitation (CPR) and Advanced Cardiovascular Life Support (ACLS) at the scene until either the heart is restarted or resuscitation efforts are considered hopeless and discontinued. An alternative strategy for those with refractory OHCA is expedited transport with ongoing mechanical CPR to an Emergency Department capable of performing extracorporeal cardiopulmonary resuscitation (ECPR). The purpose of study is to test if this strategy is feasible and beneficial.

DETAILED DESCRIPTION:
Out-of-hospital sudden cardiac arrest (OHCA) is a life-threatening condition in which the heart suddenly stops beating and there is no blood flow to the body. If cardiac arrest is not treated immediately, it causes sudden death. In the U.S. alone, over 300,000 people per year have OHCA, and less than 1 out of 10 survive. Therefore, it is important to study new ways of treating cardiac arrest patients in order to improve survival.

The current standard practice for treating OHCA is to perform CPR and Advanced Cardiovascular Life Support (ACLS) at the scene until either the heart is restarted or resuscitation efforts are considered hopeless and discontinued. This practice is supported by the fact that all currently proven CPR therapies can be delivered by paramedics in the field.

However, promising new strategies have emerged that are more feasible to initiate in the hospital. One such strategy is extracorporeal cardiopulmonary resuscitation (ECPR). ECPR requires placement of catheters in large blood vessels and connected to a machine to take over the work of the heart and lungs.

This purpose of this study is to examine the feasibility and potential benefit of expedited transport with ongoing mechanical CPR for patients with refractory OHCA patients to an Emergency Department capable of initiating ECPR.

FDA approved this study as a staged feasibility study to enroll 15 participants and submit data prior to enrolling the second 15 participants. After enrolling 15 participants, the PI chose not to pursue an amendment to enroll additional participants due to slow accrual and research restrictions related to COVID.

ELIGIBILITY:
Inclusion Criteria:

* OHCA of presumed non-traumatic etiology requiring CPR
* Predicted arrival time at ECPR-capable hospital within timeframe specified
* Witnessed arrest or initial shockable rhythm (VT or VF)
* Persistent cardiac arrest after initial cardiac rhythm analysis and shock (if shock is indicated)

Exclusion Criteria:

* Sustained return of spontaneous circulation (ROSC)
* Advanced directive indicating do not attempt resuscitation (DNAR) or do not intubate (DNI)
* Preexisting evidence of opting out of study
* Prisoner
* Pregnant (obvious or known)
* ECPR capable ED is not at the destination hospital as determined by EMS
* Legally authorized representative (LAR) or family member aware of study and refuses study participation at the scene

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Neumar, MD, PhD, Principal Investigator — University of Michigan; Robert H Bartlett, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hsu CH, Meurer WJ, Domeier R, Fowler J, Whitmore SP, Bassin BS, Gunnerson KJ, Haft JW, Lynch WR, Nallamothu BK, Havey RA, Kidwell KM, Stacey WC, Silbergleit R, Bartlett RH, Neumar RW. Extracorporeal Cardiopulmonary Resuscitation for Refractory Out-of-Hospital Cardiac Arrest (EROCA): Results of a Randomized Feasibility Trial of Expedited Out-of-Hospital Transport. Ann Emerg Med. 2021 Jul;78(1):92-101. doi: 10.1016/j.annemergmed.2020.11.011. Epub 2021 Feb 1. PMID 33541748
- See also: EROCA Study Website — https://www.medicine.umich.edu/dept/emergency-medicine/eroca-study

RESULTS

PARTICIPANT FLOW:
Groups:
- Expedited Transport: Intervention: Expedited Transport with Mechanical CPR.
  After initial Basic Life Support (BLS) and Advanced Cardiovascular Life Support (ACLS) by Emergency Medical Services (EMS) per existing EMS protocols, patients with refractory cardiac arrest are transported to an ECPR capable emergency department with ongoing mechanical CPR and ACLS for possible initiation of extracorporeal cardiopulmonary resuscitation (ECPR).
  Expedited Transport With Mechanical CPR: Patients with OHCA refractory to initial BLS and ACLS will be transported by EMS with ongoing mechanical CPR and ACLS to an emergency department capable of initiating ECPR.
Period: Overall Study
Arm/Group | Standard Care | Expedited Transport
Started | 3 | 12
Completed | 3 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care | Expedited Transport | Total
Number analyzed (Participants) | 3 | 12 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (3) | 62 (8) | 62 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 2 | 8 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 3 | 9 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Initial cardiac rythm [Count of Participants; unit: Participants]
  Ventricular fibrilation | 3 | 5 | 8
  Witnessed pulseless electrical activity (PEA) | 0 | 4 | 4
  Witnessed asystole | 0 | 3 | 3
Bystander CPR [Count of Participants; unit: Participants] | 3 | 10 | 13
Cardiac Arrest Locaion [Number; unit: participants]
  Home | 2 | 10 | 12
  Public Location | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Emergency Department Arrivals Under 30 Minutes
Description: Proportion of patients with emergency department (ED) arrival less than or equal to 30 minutes from 911 call (or cardiac arrest onset if witnessed by EMS personnel).
Time Frame: Measured within one hour cardiac arrest onset
Population: Standard care participants received EMS protocols at the scene, and thus were not included in this analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Expedited Transport
Number analyzed (Participants) | 0 | 12
Participants |  | 5

2. Primary Outcome: ECPR Initiations Under 30 Minutes
Description: Proportion of ECPR eligible patients with ECPR flow initiated less than or equal to 30 minutes from ED arrival
Time Frame: Measured within 2 hours of cardiac arrest onset
Population: Analysis includes participants eligible for ECPR.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Expedited Transport
Number analyzed (Participants) | 0 | 5
Participants |  | 3

3. Other Pre Specified Outcome: Functional Neurological Outcome: CPC
Description: Cerebral Performance Category score is widely used in cardiac arrest research to assess neurologic outcome
Time Frame: At time of hospital discharge (an average of 7 days) and 90 days after cardiac arrest
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Functional Neurological Outcome: mRS
Description: modified Rankin Score commonly used for measuring the degree of disability or dependence in the daily activities of people who have suffered a neurological disability.
Time Frame: At time of hospital discharge (an average of 7 days) and 90 days after cardiac arrest
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Neuropsychological Outcome Battery: NIH Toolbox
Description: The NIH toolbox includes cognitive testing and can be administered using an iPad
Time Frame: At time of hospital discharge (an average of 7 days) and 90 days after cardiac arrest
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Neuro Quality of Life: Neuro QoL
Description: Quality of Life in Neurological Disorders is a measurement system that evaluates and monitors the physical, mental, and social effects experienced by adults living with neurological conditions.
Time Frame: 90 days after cardiac arrest
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Safety: Composite Prevalence of 6 Specified Adverse Events
Description: Composite safety endpoint of hemorrhage requiring blood transfusion, vessel damage requiring vascular procedure or leading to occlusion, venous/arterial thromboembolism, stroke, renal failure, and infection.
Time Frame: At time of hospital discharge (an average of 7 days) and 90 days after cardiac arrest
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Participants were followed for 90 days after intervention
Arm/Group | Standard Care | Expedited Transport
All-Cause Mortality (participants affected / at risk) | 2/3 | 12/12
Serious Adverse Events (participants affected / at risk) | 2/3 | 6/12
Other Adverse Events (participants affected / at risk) | 0/3 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Care (N=3) | Expedited Transport (N=12)
Hemorrhage from cannulation site (Surgical and medical procedures) | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acute Kidney Injury (AKI) (Renal and urinary disorders) | 1 | 3
Hemorrhagic Shock (Blood and lymphatic system disorders) | 0 | 1
Hemoperitoneum (Nervous system disorders) | 0 | 1
Anoxic brain injury (Nervous system disorders) | 2 | 2
Failure to establish circuit blood flow (Cardiac disorders) | 0 | 1
Ventricular Fibrillation/Ventricular Tachycardia (Cardiac disorders) | 0 | 1
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 | 1
Cardiogenic Shock (Cardiac disorders) | 0 | 2
Acute Liver Injury (Hepatobiliary disorders) | 0 | 1
Ischemic Stroke (Nervous system disorders) | 0 | 1
Ischemic Skin Necrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Presumed Moderate Acute Respiratory Distress Syndrome (ARDS) (Reproductive system and breast disorders) | 0 | 1
Non ST Elevation Myocardial Infarction (NSTEMI) (Cardiac disorders) | 0 | 1
Tracheal aspirate - Methicillin-sensitive Staphylococcus aureus (MSSA) (Infections and infestations) | 1 | 0
Hemopericardium (Cardiac disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-15): https://cdn.clinicaltrials.gov/large-docs/47/NCT03065647/Prot_SAP_000.pdf